CLINICAL TRIAL: NCT00910936
Title: Effects of an Exercise Program on Metabolic Parameters of Patients With a HIV Infection.
Brief Title: Exercise for Patients With HIV Infections
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Fernando Dimeo, Dept. of Sports Medicine, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EA04/050/07
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: HIV Infections; Lipodystrophy; Inflammation
Keywords: HIV; Exercise; Inflammation; Quality of life; Lipodystrophia
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Inflammation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — 12 weeks endurance training, 3 times weekly for 35 minutes
  Arms: Intervention

SUMMARY:
The investigators will evaluate the effects of an endurance exercise program on the physical performance, the well being, and indicators of metabolic function in patients with an HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* HIV infection
* Antiviral therapy
* Understanding of written German

Exclusion Criteria:

* Diabetes mellitus
* All conditions which can be aggravated by exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-01 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2max) | At recruitment and after 12 weeks

SECONDARY OUTCOMES:
Quality of life | At recruitment and after 12 weeks
Indicators of fat metabolism | At recruitment and after 12 weeks
Markers of inflammation | At recruitment and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Section Sports Medicine, Charité Universitätsmedizin Berlin, Hindenburgdamm 30, Berlin, State of Berlin, Germany